CLINICAL TRIAL: NCT07301359
Title: Association of the PaO₂/PaCO₂ Ratio With ICU Mortality Independent of Oxygen Saturation and Mean Arterial Pressure: Insights From the MIMIC-II Database
Brief Title: Is the PaO₂/PaCO₂ Ratio Associated With ICU Mortality Independent of Oxygen Saturation and Mean Arterial Pressure?
Acronym: RATIO-MIMIC
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MOHAMMED FAWZI ALI ABOSAMAK, Dr. Mohammed F Abosamak 1.... Department of Anesthesia and Intensive Care Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt 2....Department of adults ICU, Security Forces Hospital Program, Central Directorate Of Medical Services , Riyadh, KSA, Tanta University
Other Study IDs: MIMIC-II
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Mortality in Intensive Care Units

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Indwelling Arterial Catheter Clinical dataset contains clinical data for 1776 patients..........: The Indwelling Arterial Catheter Clinical dataset contains clinical data for 1776 patients from the MIMIC-II clinical database. It was the basis for the article: Hsu DJ, et al. The association between indwelling arterial catheters and mortality in hemodynamically stable patients with respiratory failure: A propensity score analysis. Chest, 148(6):1470-1476, Aug. 2015.This dataset was also used by Raffa et al. in Chapter 5 "Data Analysis" of the forthcoming book: Secondary Analysis of Electronic Health Records, published by Springer in 2016......................................................................................................................................................................................................................................................................................................................................................................................................................................................................

SUMMARY:
The goal of this observational study is to learn about the Association of the PaO₂/PaCO₂ Ratio with ICU Mortality Independent of Oxygen Saturation and Mean Arterial Pressure

ELIGIBILITY:
Inclusion criteria

Adult patients (≥ 18 years old) at time of ICU admission. Rationale: Restrict to adult physiology and consent/ethics comparability.

First ICU stay during hospital admission (index ICU admission). Rationale: Avoid within-hospital dependency and repeated measures bias.

ICU admission captured in the MIMIC-II dataset between the database start and end dates.

Rationale: Use all eligible records within the dataset timeframe.

At least one arterial blood gas (ABG) measurement with both PaO₂ and PaCO₂ available during the ICU stay.

Rationale: Primary exposure is PaO₂/PaCO₂ ratio; require both values to compute it.

Available outcome data for ICU mortality (discharge status from ICU). Rationale: Necessary to ascertain primary endpoint.

Available SpO₂ and mean arterial pressure (MAP) measurements in the same ICU stay (for confounder adjustment).

Rationale: Study aims to evaluate independence from SpO₂ and MAP; require at least one measurement of each during the stay. (If either is missing, see handling below.)

Exclusion criteria

Age < 18 years. Rationale: Exclude pediatric physiology.

Missing or unusable arterial blood gas values (PaO₂ or PaCO₂ absent or non-numeric) for the ICU stay.

Rationale: Cannot compute exposure.

No recorded ICU outcome (missing ICU discharge status) or lost/invalid mortality data.

Rationale: Cannot determine primary outcome.

Extreme or physiologically implausible ABG values that suggest data error (e.g., PaO₂ ≤ 0 mmHg, PaCO₂ ≤ 0 mmHg, or PaO₂ > 1000 mmHg or PaCO₂ > 300 mmHg - thresholds may be tightened after exploratory data review).

Rationale: Remove likely data-entry errors. Document thresholds and perform sensitivity analysis.

Patients on extracorporeal life support (ECMO) during ABG measurement (if identifiable in MIMIC-II).

Rationale: ECMO profoundly alters gas exchange and PaO₂/PaCO₂ physiology; consider exclusion or separate subgroup.

Repeat ICU admissions within the same hospital stay beyond the index admission (if you choose to restrict to single index admission).

Rationale: Prevent correlated observations - include only the first ICU stay per hospital admission.

ICU stays with no recorded SpO₂ or MAP at any time (if you insist on requiring these for adjustment).

Rationale: If primary models must adjust for SpO₂ and MAP, exclude records without those covariates or plan appropriate imputation.

Do-not-resuscitate (DNR)/comfort-care only status recorded before ABG measurement (optional exclusion depending on study question).

Rationale: Treatment limitation orders can confound mortality associations; you may choose instead to adjust or analyze separately.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included adult patients admitted to intensive care units (ICUs) represented in the Medical Information Mart for Intensive Care II (MIMIC-II) database, a large, publicly available critical care database developed by the Massachusetts Institute of Technology (MIT) in collaboration with Beth Israel Deaconess Medical Center (BIDMC). The database contains detailed, de-identified clinical data from patients admitted to the BIDMC ICUs between 2001 and 2008.
  All adult (≥18 years) ICU patients with at least one arterial blood gas measurement containing both arterial oxygen tension (PaO₂) and arterial carbon dioxide tension (PaCO₂) were eligible for inclusion. For each included ICU stay, corresponding measurements of oxygen saturation (SpO₂) and mean arterial pressure (MAP) were also extracted to allow adjustment for oxygenation and hemodynamic status.
  Patients were excluded if they lacked valid PaO₂ or PaCO₂ measurements, had missing ICU mortality data, or had physiologically impla
Sampling Method: Non-Probability Sample
Enrollment: 1776 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2016-03-20 (Actual); Study Completion 2016-03-20 (Actual)

PRIMARY OUTCOMES:
ICU mortality | From October 2025 to January 2026.............................................................................................................................................................................................................................
  Death occurring during the ICU stay

SECONDARY OUTCOMES:
28-day all-cause mortality | From October 2025 to January 2026
  28-day all-cause mortality

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT07301359/Prot_SAP_000.pdf